CLINICAL TRIAL: NCT04857788
Title: Randomized Controlled Trial for Efficacy Assessment of a Program of Digital Accompaniment to Optimize Homework Performances and Increase Familial Quality of Life in 9 to 16 Years Children With ADHD" - PANDA-H
Brief Title: Program of Digital Accompaniment to Optimize Homework Performances and Increase Familial Quality of Life in 9 to 16 Years Children With ADHD
Acronym: PANDA-H
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC20_0070
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pandah Application only (Experimental): Design is a controlled randomized Study with two parallel arms after randomization with a three months follow-up of the two arms that are (Group 1) Care as usual for patients in follow-up list; (Group 2) PANDAH App proposed alone with only 15-20 minutes setup with investigator at start-up (digital accompaniment only); Patients of the 2 groups will have a three months follow-up period before secondary evaluation and entering into the so-called extension period.
  Interventions: Other: Pandah Application smartphone only
- Care as usual (No Intervention): Design is one period of 3 months with 2 parallel groups (with or without application) following by extension period of 3 months with all subject accessing to the application.

INTERVENTIONS:
Other: Pandah Application smartphone only — Patients will have an application on their smartphone to help them do their homework
  Arms: Pandah Application only

SUMMARY:
Attention Deficit Disorder with or without Hyperactivity (ADHD) is a frequent pathology in children that has important consequences on schooling both in terms of academic level (due to the attentional disorder) and behavior (disruption of the class). ADHD also has an impact on family functioning, which can generate stress and family altercations. The homework period can be a particularly tense time and a source of conflict with the child, which has negative consequences on the family atmosphere, learning efficiency and of course academic success.

The investigators wish to evaluate an innovative digital device (a smartphone application) to accompany the child during homework periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 9-16 years old with ADHD assessed by Conners 3 scales
* Parents and children giving informed consent
* Patients in follow-up list of participant centers
* Patients with unchanging care for the last 3 months (medication and therapy)

Exclusion Criteria:

* Patients with severe psychiatric disease such as schizophrenia, bipolar disorder, or autism spectrum disorders and suicidal behavior (all assessed by Child Behavior Checklist Scale)
* Patients with no smartphone or not easy access to smartphone (ie patients of social facilities, internship…)
* Patients with mild to severe mental retardation or that may obviously not be able to use the app
* Patients included in special program other the Care as Usual (defined in the ADHD French network) in follow-up list.
* Patients with Methylphenidate treatment or change of titration for less than 3 months.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare Homework Performance in the PANDAH group vs Usual Care Only group in ADHD patients at 3 months. | 3 months
  Global score of Homework Performance Questionnaire (HPQ), Parent version at 3 months. • Homework Performance Questionnaire = HPQ Parental and Teacher version are a 27 (Parental) and 25 (teacher) items scale scored form 0 (never) to 3 (very often). Total score is a sum of item's scores. Highest score is the worst. Min : 0 Max 108 (Parental) and 100 (Teacher)

SECONDARY OUTCOMES:
Change in Homework Performance assessed by Parents collected at 0, 3 and 6 months between the PANDAH group and Usual Care group | 0, 3, 6, Months
  Global score and domain scores of Homework Performance Questionnaire (HPQ), Parent version at Month 0, Months 3, and Months 6. • Homework Performance Questionnaire = HPQ Parental and Teacher version are a 27 (Parental) and 25 (teacher) items scale scored form 0 (never) to 3 (very often). Total score is a sum of item's scores. Highest score is the worst. Min : 0 Max 108 (Parental) and 100 (Teacher)
Change in Homework Performance assessed by Teachers at 0, 3 and 6 months between the PANDAH group and usual care group in ADHD patients | 0, 3 and 6 months
  Global score and domain scores of Homework Performance Questionnaire (HPQ), Teacher version at 0, 3 and 6 months. • Homework Performance Questionnaire = HPQ Parental and Teacher version are a 27 (Parental) and 25 (teacher) items scale scored form 0 (never) to 3 (very often). Total score is a sum of item's scores. Highest score is the worst. Min : 0 Max 108 (Parental) and 100 (Teacher)
Change in patient and Family Quality of Life collected at 0, 3 and 6 months between the PANDAH group and Usual Care group. | 0, 3 and 6 months
  Patient PedSQL and PedSQL Family Impact Module at 0, 3 and 6 months. • Pediatric Quality of Life Inventory, PedSQL is a 23 items scale in 4 domains (physical capacity, emotion, relationship, and school). Scored from 0(not a problem) to 4 (always a problem). Total score is a sum of item's scores. Highest score is the worst. For children and adolescent. Min O Max 115
Change in Homework Problems assessed by Parents at 0, 3 and 6 months between the PANDAH group and Usual Care group in ADHD patients. | 0, 3 and 6 months
  Global score of Homework Problem Checklist for Parents at 0, 3 and 6 months. • Homework Problem Checklist = HPC parental version is a 20 items scale scored form 0 (never) to 3 (very often). Total score is a sum of item's scores. Highest score is the worst. Min : 0 Max : 80
To evaluate patients' ADHD Core Symptoms in the PANDAH group and Usual Care group in at 0, 3 and 6 months | 0, 3 and 6 months
  Inattention and Hyperactivity score of Conners at 0, 3 and 6 months. • Conners scale for parents is a 28 items scale in 3 domains (behavioral disturbances, impulsivity / hyperactivity, and attention disorders). Scored: not at all / a little / a lot / massive (0 to 3). Total score is a sum of item's scores. Highest score is the worst. Min O Max 112
To evaluate use/compliance of PANDAH App in the PANDAH group at 6 months and on the whole academic year. | 6 months
  In-App score of filling rate and number of complete App sessions during 6 months. • In-App filling rate is the raw data from the smartphone application regarding the usage (number of interactions, duration of activity on each screen and schedule of usage). Score must be appreciated, there is no positive or negative. Scores are variable : number of interaction is O to infiny / Duration to activity is O to infiny and Schedule of usage is time and date.
To Evaluate patients' Anxiety and Depressive Symptoms in the PANDAH group and Usual Care group at 0, 3 and 6 months | 0, 3 and 6 months
  CDRS depression and Hamilton Anxiety at 0, 3 and 6 months. • Child Depression Rating Scale = CDRS is a 17 items scale exploring depression. Items are rated form 1 to 5, 1 to 6 or 1 to 7. Sum of all items make a total score. Highest score is the worst. Min O Max 108
To measure global academic efficacy in the PANDAH group and Usual Care group at 3 and 6 months, and/or according PANDAH App use intensity. | 3 and 6 months
  Lickert scale addressed to Teachers at 3 and 6 months. • Lickert scale is a analogic scale from 0 to 10 for perceived quality of homework. O is poor and 10 is excellent. Best score is the highest score. Min 0 Max 10

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Berquin, Amiens
  - Bioulac, Bordeaux
  - Fourneret, Lyon
  - Purpuer, Montpellier
  - Olivier Bonnot, Nantes
  - Caci, Nice
  - Delorme, Paris
  - Schroder, Strasbourg
  - Speranza, Versailles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gollier-Briant F, Ollivier L, Joalland PH, Mouchabac S, Leray P, Bonnot O. Digital Homework Support Program for Children and Adolescents With Attention-Deficit/Hyperactivity Disorder: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Nov 21;13:e44553. doi: 10.2196/44553. PMID 39571155